CLINICAL TRIAL: NCT01809717
Title: Modulating The Toxicity And Efficacy Of High Dose Chemotherapy For Multiple Myeloma Through An Intervention To Increase Lean Body Mass
Brief Title: Multiple Myeloma and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 13412
Record Dates: First submitted 2013-03-05; First posted 2013-03-13 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Newly Diagnosed Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weight Lifting Exercises (Experimental)
  Interventions: Other: Weight Lifting Exercises

INTERVENTIONS:
Other: Weight Lifting Exercises

SUMMARY:
This study will establich the feasibility of weight lifting exercise among patients with multiple myeloma, determine if weight lifting exercise increases lean body mass among patients with multiple myeloma and obtain further preliminary data on toxicity and pharmacokinetics of high-dose melphalan.

DETAILED DESCRIPTION:
This is a prospective, single-institution, pilot study of a 3 month weight lifting program designed to increase musle hypertrophy prior to starting stem cell collection and receiving high-dose melphalan, in patients with multiple myeloma. We will use this exercise intervention while patients are receiving initial induction chemotherapy in the 3-6 month period before they receiv high-dose melphalan. The primary study endpoint is to determine the feasibility of recruiting and retaining multiple myeloma patients to an exercise intervention trial. The secondary study endpoint is to determine whether the weight lifting program increases lean body mass as intended.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed multiple myeloma
* 1 year since start of treatment for myeloma
* Patient and treating physician in agreement to proceed with autologous transplant, with a planned time betwwen study enrollment and transplant of 10 weeks
* Age 18 years.
* Able to walk for 6 minutes unaided.
* Body mass index 50 kg/m2
* Serum creatinine 2.5 mg/dL
* Ability to understand the informed consent document and willingness to consent. Written informed consent must be obtained from all patients before study entry.

Exclusion Criteria:

* Recent (in the past 6 months) participation in progressive weight lifting exercises or who already exercise regulary (3 times a week of moderate intensity aerobic exercise).
* Plan to move out of the area during the study intervention.
* A psychological, social, or logistical barrier that the principal investigators feel would preclude completion of the study protocol.
* Plan for use of any anti-myeloma treatment other than melphalan (the use of total body irradiation will NOT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, Principal Investigator — Abramson CC
Locations (1):
- Abramson Cancer Center of the Unviersity of Pennsylvania, Philadelphia, Pennsylvania, United States